CLINICAL TRIAL: NCT06720194
Title: Upper-limb Functional Recovery With Virtual Reality System (BTs-Nirvana) Associated With Conventional Therapy in Hospitalized Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lorena Aguilar Cano (Other)
Collaborators: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor-Investigator, Lorena Aguilar Cano, Principal Investigator, Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Organization: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RVACV2020
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Subacute Stroke
Keywords: stroke rehabilitation; upper limb recovery; physical therapy; virtual reality therapy; daily-life activities; randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This arm receives the virtual therapy plus the usual treatment
  Interventions: Device: Virtual therapy
- Control Group (Other): This arm receives the usual treatment at the same dose and time than experimental group
  Interventions: Other: Usual treatment

INTERVENTIONS:
Device: Virtual therapy — Virtual therapy has been applied for four weeks, three times a week. We administered a total of twelve sessions with a duration of 30 minutes each. Prior to virtual therapy experimental group have received kinesitherapy for 15 minutes to improve and prevent muscle spasticity and joint contractures. Therapists recorded the order of the session and they have providen the same external aid to all patients. Two days a week the experimental group have received the conventional treatment for 45 minutes (kinesitherapy, strengthening exercises muscle, trunk control, transfers, standing and walking). In addition to physiotherapy treatment, participants have done occupational therapy 5 days a week (training to perform ADLs, tracking techniques and search, manipulation, reach and grasping of different utensils, etc.), for 30 minutes each session.
  Arms: Experimental group
Other: Usual treatment — Patients assigned to the control group have received the conventional treatment five days a week. They have done physiotherapy session and occupational therapy for 45 and 30 minutes a day each one.
  Arms: Control Group

SUMMARY:
The goal of this pilot study is to evaluate if a semi-inmersive virtual reality device works in the recovery of the function of the upper limb affected in hospitalized patients who have suffered a stroke.

Reseachers will compare the virtual reality device plus the usual treatment to usual treatment to see if virtual reality device works to recovery upper limb function.

Participants will be able to receive conventional treatment or virtual therapy plus conventional treatment 5 days a week for 4 weeks.

When they are discharged, they will come to the hospital 2 times to be reviewed, 3 months and 1 year after receiving treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke confirmed by neuroimaging.
* No previous stroke.
* Subacute phase (between 1 and 6 months after the stroke).
* Ability to sit with or without support.
* Maximum 4 on the Muscle Strength Scale (MRC) for shoulder flexion and flexion-extension of the elbow of the upper limb on the affected side.
* Ability to understand and accept study procedures and to sign an informed consent having been previously informed.

Exclusion Criteria:

* Previous history of brain injury, stroke and neurological or neuropsychiatric diseases.
* Cognitive alterations, dementia, aphasia or other alteration that causes inability to understand the meaning of the study.
* Clinical inestability
* Loss of visual capacity that difficults recognizing figures on the screen.
* Orthopedic conditions involving upper limbs.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Upper limb motor function as assessed by Fugl-Meyer Upper-Limb scale (FM-UL) | at baseline, 4 weeks, 3 months and a year after treatment
  The maximum value of the motor function in the FM-UL scale is 66 points. A higher score corresponds to a better state of operation of the patient.

SECONDARY OUTCOMES:
Daily-life activities as assessed as Barthel Index (BI) | at baseline, 4 weeks, 3 months and a year after treatment
  BI evaluates 10 daily-life activities: eating, wash, dress, groom, defecate, urinate, go to the toilet, move, chair-bed, ambulation, going up and down stairs. The total score ranges from 0 to 100. The global results are grouped into four categories of dependency: total, severe, moderate or mild. Lower score means subject has more dependence ant higher score means more independence.
Trunk control as assessed as Control Trunk Test (TCT) | at baseline, 4 weeks, 3 months and a year after treatment
  TCT is a simple test that explores four movements. Each of the sections are scored as follows: 0 points if the patient is unable to perform the movement without assistance, 12 points if able to perform the movement abnormally and 25 points if the patient is able to complete the movement normally. The total score is the sum of the results of the four tests and its value can range from 0 to 100.
Daily-life activities as assessed as Self-Assessment of Role Performance and Activities of Daily Living (SARA-TM) | at baseline, 4 weeks, 3 months and a year after treatment
  SARA-TM is a questionnaire that users fill out with the orientation of the therapists. It is based on their perceptions of various daily-life activities. We have asked about items related to self-care, food, maintenance of postures, movement, manipulation and pain. Each one of the domains consists of different items that correspond to different activities. Each item is scored from 0 to 4 depending on the degree of difficulty in performing the activities. Lower values represent better function

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Regional de Malaga, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No